CLINICAL TRIAL: NCT02540304
Title: Teen Pregnancy Prevention Replication Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abt Associates (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Decision Information Resources (DIR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HHSP23320095624WC
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Teen Pregnancy; Sexual Risk-taking Behaviors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TPP program (Experimental): Reducing the Risk, Safer Sex Intervention, Cuidate!
  Interventions: Behavioral: Reducing the Risk
- Business as Usual (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Reducing the Risk — Safer Sex is a clinic-based intervention intended to reduce the incidence of STIs and increase condom use among high-risk sexually active female adolescents and delivered in face-to-face individualized sessions by a female health educator. Reducing the Risk is a sexuality-education curriculum, most often delivered in a school setting that provides instruction and practice in the social skills needed to put into action what students learn about preventing pregnancy and reducing unsafe behavior in future high-risk situations. ¡Cuidate! is adapted from the Be Proud! Be Responsible! curriculum and culturally tailored for Latino youth. It aims to reduce HIV risk and unintended pregnancies by affecting sexual behaviors such as intercourse, number of partners, and condom use.
  Other Names: Safer Sex Intervention; Cuidate!
  Arms: TPP program

SUMMARY:
This study is evaluating the effectiveness of three evidence-based teen pregnancy prevention (TPP) programs in reducing sexual risk-taking behaviors of youth. The study is using an experimental design in which youth are randomly assigned to receive either TPP programming or services as usual.

DETAILED DESCRIPTION:
The Teen Pregnancy Prevention Replication Study is being conducted under contract for the U.S. Department of Health and Human Services (DHHS) Office of the Assistant Secretary for Planning and Evaluation (ASPE) and Office of Adolescent Health (OAH) by Abt Associates and its subcontractors, Belmont Research Associates, and Decision Information Resources (DIR). The study seeks to add to the knowledge base about effective teen pregnancy prevention programs by examining replications of evidence-based program models currently funded through the Teen Pregnancy Prevention program, administered by OAH.

Through a series of rigorous experimental design evaluations, the study will test multiple replications of three widely-used evidence-based program models to determine their effectiveness across different settings and populations. This strategy of selecting multiple replications of each program model will allow for an examination of variation in impacts across replications for each program model and provide evidence about the generalizability of program effectiveness. A comprehensive implementation study will provide information about the contexts in which evidence-based programs are implemented, the challenges faced in implementing them, and the aspects of program implementation that are associated with program impacts.

The models that will be examined in this study include: ¡Cuidate! (an HIV/STI risk reduction program); Reducing the Risk (a sexuality education curriculum); and Safer Sex (a clinic-based HIV/STI prevention program for high-risk adolescent females). Program impacts will be estimated by using an experimental design in which youth are randomly assigned to treatment and control conditions. The unit of random assignment will be the individual or school class, depending upon the program setting.

Overall, the study will be based on a sample of approximately 8,000 youth in nine locations across the country. The evaluation team will collect baseline information when youth are enrolled in the program, short-term outcome data at a follow-up survey between 6 and 12 months post-random assignment, and longer-term outcome data at a follow-up survey administered between 18 and 24 months post-random assignment. Comparison of outcomes for program and control groups will provide important information about the effectiveness of the programs in reducing teen pregnancy and associated risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* youth at risk active consent parent permission

Exclusion Criteria:

-

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7620 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sexual activity in the last 90 days | 6 months after baseline
  single dichotomous outcome on self-report questionnaire
Sexual Risk in the last 90 days | 6 months after baseline
  single dichotomous outcome on self-report questionnaire

SECONDARY OUTCOMES:
Use of Birth Control in the last 90 days | 6 months after baseline
  single dichotomous outcome on self-report questionnaire
Knowledge of Sexually transmitted infections | 6 months after baseline
  Average of 12 dichotomous items on self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Meredith C Kelsey, PhD, Principal Investigator — Abt Associates Inc